CLINICAL TRIAL: NCT04820244
Title: Characterizing Rate of Progression in USHer Syndrome (CRUSH) Study
Acronym: CRUSH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Ushersyndroom (Unknown)
Responsible Party: Sponsor
Other Study IDs: NL67258.091.18
Record Dates: First submitted 2021-03-01; First posted 2021-03-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Usher Syndrome, Type 2A; Retinitis Pigmentosa; USH2A
Keywords: USH2A; Non-Syndromal USH2 related Retinitis Pigmentosa; Natural history study
MeSH Terms: conditions — Usher syndrome, type 2A; Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- No intervention: Otherwise healthy human volunteers, 16-55 years old, with a confirmed genetic diagnosis of Usher Syndrome type 2 or non-syndromal USH2A related retinitis pigmentosa
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Mutations in USH2A give rise to two phenotypes: Usher syndrome type 2a (USH2A) and nonsyndromic RP (USH2A associated nsRP). Usher syndrome is the most common form of congenital deafblindness. Patients with Usher syndrome are hearing impaired or profoundly deaf from birth and this can be rehabilitated with hearing aids or a cochlear implant. Furthermore, these patients develop retinitis pigmentosa (RP), a slowly progressive type of retinal degeneration that usually starts in the first or second decade of life. In both USH2A and nsRP patients the disease leads to severe visual impairment and eventually blindness around the 50th-70th year of life. There are no treatment options for the retinal degeneration. We do not know if they also suffer from balance complaints.

Currently, genetic therapy for Usher syndrome type 2 and USH2A associated nsRP is in development. But to measure the effect of a (genetic) therapy, it is crucial to know the detailed natural course of the visual and hearing deterioration over time. Several genetic therapy studies for other disorders are currently delayed, because the natural history of the disease has not been studied in detail previously.

The main objective is to map the natural course of the visual and hearing deterioration in Usher Syndrome 2 and USH2A associated nsRP for upcoming genetic therapy studies. Secondary objectives are: 1) To determine the necessary type of (combined) examinations, the sample size and length of studies (in years) essential to evaluate future genetic therapy in Usher syndrome. 2) To improve counselling of patients with Usher syndrome type 2 and USH2A associated nsRP with detailed information on the prognosis. 3) To identify additional etiological factors that explain variability in hearing impairment by adding questionnaires and psychophysical audiometric tests; and to assess the vestibular phenotype in Usher syndrome type 2 and USH2A associated nsRP patients.

This is a longitudinal, prospective natural history study. The study population consists of healthy human volunteers, 16 - 55 yr old with a confirmed genetic diagnosis of Usher Syndrome type 2 or and USH2A associated nsRP.

The main study endpoint is the natural course of the visual and hearing deterioration in Usher Syndrome type 2 and USH2A associated nsRP, over a time span of 4 years.

There are no risks associated with participation.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed with rod-cone degeneration and at least two; pathogenic or likely pathogenic mutations in one of the Usher type 2 genes;
* Willing and able to complete the informed consent process;
* Ability to return for all study visits over 48 months;
* Age ≥ 16 years.

Both eyes must meet all of the following:

* Clinical diagnosis of a rod-cone degeneration;
* Clear ocular media and adequate pupil dilation to permit good quality photographic imaging;
* Ability to perform kinetic and static perimetry reliably;
* Baseline visual acuity ETDRS letter score of 54 or more [approximate Snellen equivalent 20/80 or better];
* Stable fixation;
* Clinically determined [on Octopus 900 Pro] kinetic visual field III4e area 7,5°, or more in the study eye.

Exclusion Criteria:

* Mutations in genes that cause autosomal dominant RP, X-linked RP, or presence of biallelic mutations in autosomal recessive RP/retinal dystrophy genes other than Usher genes;
* Expected to enter experimental treatment trial at any time during this study History of more than 1 year of cumulative treatment, at any time, with an agent associated with pigmentary retinopathy (including hydroxychloroquine, chloroquine, thioridazine, and deferoxamine).

If either eye has any of the following, the patient is not eligible:

* Current vitreous hemorrhage;
* Current or any history of rhegmatogenous retinal detachment;
* Current or any history of (e.g., prior to cataract or refractive surgery) spherical equivalent of the refractive error worse than -8 Diopters of myopia;
* History of intraocular surgery (e.g., cataract surgery, vitrectomy, penetrating keratoplasty, or LASIK) within the last 3 months;
* Current or any history of confirmed diagnosis of glaucoma (e.g., based on glaucoma visual field, nerve changes, or glaucoma filtering surgery);
* Current or any history of retinal vascular occlusion or proliferative diabetic retinopathy;
* Expected to have cataract removal surgery during the study;
* History or current evidence of ocular disease that, in the opinion of the investigator, may confound assessment of visual function;
* History of treatment for retinitis pigmentosa that could affect the progression of retinal degeneration (including participation in a clinical trial within the last year or a retained drug delivery device).

If either ear has any of the following, the patient is not eligible:

* The audiometric PTA(1-2-4kHz) for the best hearing ear should not exceed 75dB HL;
* Patients with bilateral cochlear implants cannot participate in the study;
* A planned, second, cochlear implantation during the study.

Ages: 16 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The Dutch Usher syndrome population consists of an estimated 850 patients. Additionally we would like to include patients with USH2A associated nsRP. Subjects will be recruited from this population. In the past years it has been clear that patients are highly motivated to participate in research for their disease. We aim to include 50 subjects and given our past experiences, we consider this a feasible number of participants. The study population consists of both males and females between 16 and 55 years of age with a confirmed genetic diagnosis of USH2A associated RP either syndromic or nonsyndromic.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2024-03-02 (Estimated); Study Completion 2024-03-02 (Estimated)

PRIMARY OUTCOMES:
Change in perceived visual functioning | Baseline, 2 years and study completion at 4 years
  Measured by the Visual Functioning Questionnaire-48 (VFQ-48): score of difficulty of performing 48 activities (items). The score is determined using two formulas: 'average item score = total item scores / (48 - U)' in which activities for which a person has non-visual reasons not to do it or in which they are not interested are scored with 'U', and '0.9*LN((2.34-average item score) / (average item score+2.22))+0.05'. The higher the score, the lower the perceived visual functioning.
Change in perceived handicap due to hearing impairment | Baseline, 2 years and study completion at 4 years
  Measured by the Speech, Spatial and Qualities of Hearing Scale (SSQ): range 0-500, the higher the score, the fewer the perceived handicap due to hearing impairment.
Change in perceived handicap due to dizziness | Baseline, 2 years and study completion at 4 years
  Measured by the Dizziness Handicap Inventory (DHI): range 0-100, the higher the score, the greater the perceived handicap due to dizziness.1. Pure tone audiometry and speech audiometry
Change in lifestyle adjustment due to Usher syndrome. | Baseline, 2 years and study completion at 4 years
  Measured by the Usher lifestyle survey: qualitative questionnaire, no quantitative measures
Change in perceived health | Baseline, 2 years and study completion at 4 years
  Measured by the 12-item Short-Form Health Survey (SF-12): 12 items with ranges 3-6, transformation of scores: ((patient score - lowest possible score)/range of scores)) * 100, the higher the score, the greater the perceived health.
Change in the indication of depressive symptoms | Baseline, 2 years and study completion at 4 years
  Measured by the Patient Health Questionnaire Mood Scale (PHQ-9): range 0-27, the higher the score, the greater the indication of depressive symptoms.
Change in overall condition of the eye | Baseline and every year until study completion at 4 years
  Measured by full ophthalmic exam.
Change in visual acuity | Baseline and every year until study completion at 4 years
  Measured by best-corrected visual acuity.
Change in visual fields area | Baseline and study completion at 4 years
  Measured by dynamic perimetry with topographical analysis.
Change in visual fields sensitivity | Baseline and every year until study completion at 4 years
  Measured by static perimetry with topographical analysis.
Change in mean retinal sensitivity | Baseline and every year until study completion at 4 years
  Measured by fundus-guided microperimetry.
Change in ellipsoid zone (EZ) area | Baseline and every year until study completion at 4 years
  Measured by optical coherence tomography (SD-OCT).
Change in retinal autofluorescence and Robson ring size | Baseline and every year until study completion at 4 years
  Measured by fundus autofluorescence imaging.
Change in condition of the retina, macula, optic nerve and ocular vascularization | Baseline and every year until study completion at 4 years
  Measured by assessing stereo color fundus photography.
Change in rod- and cone-mediated retinal function | Baseline and every year until study completion at 4 years
  Measured by full-field stimulus testing (FST).
Change in retinal function | Baseline and study completion at 4 years
  Measured by full field electroretinogram amplitudes and timing in response to rod- and cone-specific stimuli.
Change in hearing thresholds | Baseline and study completion at 4 years
  Measured by pure tone audiometry (PTA) and speech audiometry.
Change in auditory speech recognition abilities in noise | Baseline and study completion at 4 years
  Measured by the digits in noise test (DIN).
Change in integrity of the outer hair cells | Baseline and study completion at 4 years
  Measured by otoacoustic emissions (OAEs).
Change in integrity of the inner hair cells, the synapse and the first stage on the auditory nerve | Baseline and study completion at 4 years
  Measured by electrocochleography (ECochG).
Vestibular function | 3 years
  Measured by rotational chair test and calorisation.
Function of individual vestibular semicircular canals | 3 years
  Measured by video head impulse test (HIT) test.
Function of saccule and utricule of the vestibular organ | 3 years
  Measured by vestibular evoked myogenic potential (VEMP) test.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Pennings, Dr, Study Director — Radboud Universitair Medisch Centrum; Erwin van Wyk, Dr, Principal Investigator — Radboud Universitair Medisch Centrum; Carel Hoyng, Prof, Principal Investigator — Radboud Universitair Medisch Centrum; Ronald Pennings, Dr, Principal Investigator — Radboud Universitair Medisch Centrum
Locations (1):
- Radboud universitair medisch centrum, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided